CLINICAL TRIAL: NCT01934491
Title: A Novel Cognitive Training Intervention for Major Depressive Disorder
Brief Title: Cognitive Training for Depression II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 12-0266; 1K23MH099223-01 (NIH)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Major Depressive Disorder
Keywords: Cognitive training; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training A (Experimental): emotional memory training exercise
  Interventions: Behavioral: Cognitive Training A
- Cognitive Training B (Active Comparator): memory training exercise
  Interventions: Behavioral: Cognitive Training B

INTERVENTIONS:
Behavioral: Cognitive Training A
  Arms: Cognitive Training A
Behavioral: Cognitive Training B
  Arms: Cognitive Training B

SUMMARY:
This study is evaluating the effects of two brain training exercises on: memory, cognitive processing and depression symptoms.

DETAILED DESCRIPTION:
There is an urgent public health need to develop more effective and well tolerated treatments for patients with major depressive disorder (MDD); cognitive training interventions aiming to modify cognitive and affective processing abnormalities underlying MDD represent a promising new strategy. This research project translates a well established cognitive bias in major MDD, working memory bias, into a novel intervention target. In a double-blind, randomized, controlled study, MDD participants undergo 6 weeks of cognitive training sessions, with three sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* Primary, current Axis I diagnosis of Major Depressive Disorder according to DSM-IV criteria and Ham-D-17 score between 16-27
* Age 18-55
* Able to give informed consent

Exclusion Criteria:

* A history of drug or alcohol abuse or dependence (DSM-IV criteria) within 6 months
* Visual impairment that would affect the ability to observe the computerized presentation of faces.
* Motor impairment that would affect the ability to provide a response by quickly pressing a button.
* Lifetime history of Bipolar spectrum disorders or schizophrenia spectrum disorders.
* Primary, current Axis I diagnosis other than Major Depressive Disorder
* Primary, current Axis II personality disorder.
* Currently attending a cognitive-behavioral psychotherapy regimen
* Acute suicidal or homicidal risk (evidenced by suicidal or homicidal attempt within 6 months of screening)
* Pregnancy in women. Pregnant women are excluded from the study because research has shown that hormonal changes that occur during pregnancy can mimic and/or influence symptoms of depression. Including patterns of mood and cognition. These mood and cognitive changes could mask the effect of the cognitive training in this study, so pregnant women will be excluded for that reason.
* Enrolled participants can be currently taking medication but must be stabilized on their medication regimens before enrolling in the study (i.e., no medication has been started within 8 weeks, stopped within 6 weeks or titrated up or down within 4 weeks of study entry). Accordingly, if a patient's medication status must change during the course of the study, we will discontinue them in the study. We do not anticipate that this will occur frequently, as again, patients' medication regimens must be stable before enrolling in the study. No medications will be discontinued for the purpose of enrollment into the study.

Subjects must exhibit no or only moderate alcohol use. Subjects with current excessive use of alcohol (> 8 ounces/day for men and > 6 ounces/day for women) are ineligible for participation, as such drug use could confound the results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08; Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (Ham-D) | baseline and week 6
  Depression symptom severity comparison at week 6 to baseline

SECONDARY OUTCOMES:
Negative Affective Bias | baseline
  scale using Self-referential Information Processing Task; Affective Go/No-Go; Emotional Stroop
Negative Affective Bias | week 3
  scale using Self-referential Information Processing Task; Affective Go/No-Go; Emotional Stroop
Negative Affective Bias | week 6
  scale using Self-referential Information Processing Task; Affective Go/No-Go; Emotional Stroop
Working Memory | baseline
  Neurocognition
Working Memory | week 3
  Neurocognition
Working Memory | week 6
  Neurocognition

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Iacoviello, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States